CLINICAL TRIAL: NCT06737159
Title: Utility of Severity Scales in Clinical Practice in Children Hospitalized Due to Bronchiolitis: Prospective Multicentre Cohort Study.
Brief Title: Utility of Severity Scales in Clinical Practice in Children Hospitalized Due to Bronchiolitis.
Status: Not yet recruiting | Type: Observational
Sponsor: Szpital im. Św. Jadwigi Śląskiej (Other)
Responsible Party: Sponsor
Other Study IDs: 4/PNDR/2023
Record Dates: First submitted 2024-11-27; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Bronchiolitis
Keywords: bronchiolitis; bronchiolitis severity scoring; validation; utility
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Prospective observational study of patients hospitalized with bronchiolitis. The objective of our study is to compare the accuracy of commonly used clinical scales for bronchiolitis to predict relevant outcomes.

ELIGIBILITY:
Inclusion Criteria:

Children eligible for the trial must fulfil all of the following criteria:

1. Children admitted to the hospital with the clinical diagnosis of acute bronchiolitis, which is defined as an apparent viral respiratory tract infection associated with airway obstruction manifested by at least one of following symptoms:

* Tachypnoea (WHO definition).
* Increased respiratory effort manifested as follows:

  1. Nasal flaring;
  2. Grunting;
  3. Use of accessory muscles;
  4. Intercostal and/or subcostal chest wall retractions;
  5. Apnoe.
* Crackles and/or wheezing. 2. Aged 5 weeks - 24 months old.

Exclusion Criteria:

1. Diagnosis or suspicion of asthma.

Ages: 5 Weeks to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Hospitalized patients with diagnosis of bronchiolitis
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants requiring oxygen supplementation | From admission to hospital discharge up to 2 weeks
Duration of oxygen supplementation | From admission to hospital discharge up to 2 weeks
  among those requiring oxygen
The time until the infant will be assessed as being 'fit for discharge' | From admission to hospital discharge up to 2 weeks
  which is defined as the point at which the infant will be feeding adequately (taking >75% of their usual intake based on parents' assessment) and will have a saturation of at least 92% for 6 h on room air, while the axillary body temperature will remain
Worsening of clinical status, including the following | From admission to hospital discharge up to 2 weeks
  PICU admission
Adverse events, especially incidence of pneumonia | From admission to hospital discharge up to 2 weeks
  which is defined as:
  * temperature increase (fever >38 )
  * deterioration of general condition
  * inflammatory changes in lung ultrasound or chest X-ray
Hospital length of stay | From admission to hospital discharge up to 2 weeks
  (> 3 days)

CONTACTS AND LOCATIONS:
Locations (1):
- Szpital im. Św. Jadwigi Śląskiej, Trzebnica, Poland

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and/or generated during this study will be made available after the publication of results
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Avaliable after the publication
Access Criteria: Upon researcher's personal request